CLINICAL TRIAL: NCT04748783
Title: Antiviral Efficacy and Acceptability of Therapeutic Antiseptic Mouth Rinses for Inactivation of COVID SARS-2 Virus
Brief Title: Antiviral Efficacy and Acceptability of Mouth Rinses for Inactivation of COVID-19
Acronym: COL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-3046; COL Study (Other: GO Health Center)
Record Dates: First submitted 2021-02-09; First posted 2021-02-10 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2021-04

CONDITIONS: COVID19; Coronavirus Infection; SARS CoV-2 Infection
Keywords: Inactivation of SARS CoV-2 Virus; Antiseptic Mouth Rinses
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Water; Hydrogen Peroxide; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind prospective trial to test the efficacy and acceptability of 4 therapeutic, antiseptic mouth rinses to inactivate SARS-CoV-2 virus in saliva of COVID-19 positive patients
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Sterile water (Placebo Comparator): Subject participants will rinse mouth one time for 60 seconds with 10 mL of sterile water
  Interventions: Other: Water
- Peroxyl (Active Comparator): Subject participants will rinse mouth one time for 60 seconds with 10 mL Peroxyl (1.5% w/v hydrogen peroxide) rinse
  Interventions: Other: Peroxyl
- Periogard (Active Comparator): Subject participants will rinse mouth one time for 60 seconds with 10 mL Periogard (0.12% Chlorhexidine Gluconate) rinse.
  Interventions: Drug: Periogard
- Peroxyl & Periogard (Active Comparator): Subject participants will complete an on-label sequential rinse starting with Peroxyl (1st) 10ml for 60 seconds and then Periogard (2nd) 15ml for 30 seconds.
  Interventions: Other: Peroxyl; Drug: Periogard
- Colgate Total Zero (Active Comparator): Subject participants will rinse mouth one time with Colgate Total Zero Fresh Breath (0.075% Cetylpyridinium Chloride) 20ml for 30 seconds
  Interventions: Other: Colgate Total Zero

INTERVENTIONS:
Other: Water — Subject participants will rinse mouth one time for 60 seconds with 10 mL of sterile water.
  Other Names: Sterile Water
  Arms: Sterile water
Other: Peroxyl — Subject participants will rinse mouth one time for 60 seconds with 10 mL Peroxyl (1.5% w/v hydrogen peroxide) rinse
  Other Names: Colgate® Peroxyl® Mouth Sore Rinse
  Arms: Peroxyl; Peroxyl & Periogard
Drug: Periogard — Subject participants will rinse mouth one time for 60 seconds with 10 mL Periogard (0.12% Chlorhexidine Gluconate) rinse.
  Other Names: Colgate® PerioGard® Rinse
  Arms: Periogard; Peroxyl & Periogard
Other: Colgate Total Zero — Subject participants will rinse mouth one time with Colgate Total Zero Fresh Breath (0.075% Cetylpyridinium Chloride) 20ml for 30 seconds
  Other Names: Colgate Total® Mouthwash
  Arms: Colgate Total Zero

SUMMARY:
Subjects (125) will be randomized to one of five mouthrinses and will be asked to give a saliva sample immediately before and after a 30-60 second mouthwash.

Saliva samples will be collected from subjects at 15-minute intervals thereafter up to one hour (15, 30, 45 and 60 min). The saliva will be used for RT-PCR detection of Severe Acute Respiratory Syndrome CoronaVirus 2 (SARS-CoV-2) and viral infectivity assays, along with quantitative cytokine and chemokine concentration (pg/mL, Luminex).

Subjects will complete a short survey on the taste and experience of using the mouthwash.

Peripheral blood will be collected at the end of salivary collection. Subjects, except controls, will be provided materials and oral hygiene instruction related to daily use of oral hygiene products. In the seven-day period between study visit one and study visit two, subjects will be directed to brush with Colgate toothpaste (at least twice per day) and rinse with the Colgate mouthrinse (according to on-label procedures). Controls are asked to carry out their typical oral hygiene regimen with the products they typically use.

All subjects keep a daily diary of oral hygiene performance, product usage, COVID-19 symptoms and exposures. Subjects complete study visit two one week after the baseline visit during which additional salivary (1 time point, 2 mL of saliva over 5 min, no rinse) will occur and blood samples collected. each subject will undergo a periodontal exam.

DETAILED DESCRIPTION:
Randomized, double-blind prospective trial to test the efficacy and acceptability of therapeutic, antiseptic mouth rinses to inactivate SARS-CoV-2 virus in saliva of SARS-CoV-2+ patients 18-65 years of age. The study will enroll 30 outpatient SARS-CoV-2+ subjects per mouth rinse, (to achieve a total of 25 subjects with full data sets per mouth rinse,) with 5 mouth rinses, requiring us to enroll 125 SARS-CoV-2+ patients. Patients will be randomized to their mouthrinse. These patients will have already had a confirmed SARS-CoV-2+ test prior to enrollment. There will be no stratification to our randomization. All mouthrinses are commercially available Colgate products and will be used according to on-label instructions.

Subjects will be randomized to a mouthrinse and will be asked to give a saliva sample immediately before and after a 30-60 second mouthwash.

Saliva samples will be collected from subjects at 15-minute intervals thereafter up to one hour (15, 30, 45 and 60 min). The saliva samples will be stored and used for RT-PCR detection of SARS-CoV-2 virus and viral infectivity assays, along with quantitative cytokine and chemokine concentration (pg/mL, Luminex).

Subjects will also complete a short survey on the taste and experience of using the mouthwash.

Peripheral blood will be collected at the end of salivary collection. Subjects, except controls, will be provided materials and oral hygiene instruction related to daily use of oral hygiene products provided by the study. In the seven-day period between study visits, subjects will be directed to brush with Colgate toothpaste (at least twice per day) and rinse with the Colgate mouthrinse (according to on-label procedures). Controls are not given Colgate products and will be asked to carry out their typical oral hygiene regimen with the products they typically use. All subjects will be asked to keep a daily diary of oral hygiene performance, product usage, COVID-19 symptoms and exposures.

Subjects will be scheduled to return to the research clinic at one week after the baseline assessment, during which additional salivary (1 time point, 2 mL of saliva over 5 min, no rinse will occur) and blood samples will be collected. At the conclusion of sample collection, the subject will undergo a periodontal exam. Study participation concludes following the periodontal exam at the end of the second on site study visit. Patients with any periodontitis or gingivitis diagnosis will be informed of their diagnosis and will be referred to an oral healthcare provider for further treatment. This study involves two 90-minute visits.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

* Diagnosed SARS-CoV-2+ status. Either became symptomatic in the prior 7 days, or if not symptomatic, likely infected/exposed within the prior 7 days. All patients listed from the University of North Carolina at Chapel Hill (UNC) Respiratory Diagnostic Center (RDC) have a confirmed SARS-CoV-2 infection and have consented to be contacted for research purposes. For patients contacting study coordinators for enrollment, who were not tested in the RDC, they must provide written proof of positive SARS-CoV-2 status in the prior 7 days.
* Individuals (all sex, all gender) at least 18 years of age and at most 65 years of age and in good oral health without any known allergies to commercial dental products or cosmetics. American Society of Anaesthesiologists (ASA) class I or II prior to SARS-CoV-2 infection.
* Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial and all of their questions have been answered.
* Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based on research site personnel's assessment.
* Females of childbearing potential will have a negative urine pregnancy test (on site) or be physically incapable of pregnancy (implants or injections, Intrauterine device, Bilateral tubal ligation, Hysterectomy, Ovariectomy, Women post-menopausal)

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* Patients who have been eating or drinking within an hour of the study
* Patients under 18 years of age and older than 65 years of age
* Subjects presenting with and/or self-reporting any of the following will not be included in the study:

  * history of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses. (self-reported)
  * Self-reported allergy to hydrogen peroxide, peroxyl, chlorhexidine gluconate, periogard, peridex, colgate total zero, colgate total, cetylpyridinium chloride, essential oils (Eucalyptol, Menthol, Methyl salicylate, Thymol), and other components in the mouth rinses (methyl salicylate, ethanol, saccharin sodium, glycerin, propylene glycol, sorbitol, Federal Food, Drug, and Cosmetic (FD&C) blue additive no. 1, Poloxamer 407, Benzoic acid, Zinc chloride, Sodium benzoate, Sucralose, Polyethylene Glycol (PEG-40) sorbitan diisostearate, potassium sorbate, citric acid).
  * History of serious medical conditions that, at the discretion of the Investigator, will disqualify the subject. (Self-reported)
  * A history of severe dry mouth (xerostomia), severe drug-induced xerostomia (antidepressants, anticonvulsants, antihypertensives), or Sjogren's syndrome
  * A history of recent (within the last 30 days) or current recent oral herpes flare up, candida (thrush) infection, apthous ulcer flare up, current/active severe periodontal disease, or other recent oral viral infection or flare up within the past 30 days (self-reported)
  * Current history of alcohol or drug abuse (self-reported).
  * History of drinking water or eating food within an hour of the study visit.
  * History of drinking alcohol within 12 hours of the study visit.
  * History of using a commercial mouthrinse within 24 hours of the study visit.
  * Participation in any study involving oral care products, concurrently or within the previous 30 days. (self-reported)
  * Positive pregnancy test reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results. Additionally, women are advised to check with their physician before using Chlorhexidine Gluconate during pregnancy and lactation, which cannot occur in a blinded, randomized trial.)
  * Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this trial.
  * Patient with developmental/cognitive disability that cannot self-consent, comprehend and follow the requirements of the study based on research site personnel's assessment.
  * Patients with sizable mucosal tears, abrasions, growths or burns in the mouth
  * Patients with kidney dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura a Jacox, DMD, PhD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Adams School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning following publication up to 1 year provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Following publication up to 1 year
Access Criteria: Investigator who proposes to use the data has approval from an IRB, IEC, or REB as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] State Officials Announce Latest COVID-19 Facts Including New Data on Racial Demographics and Expanded Health Care Worker Data. California Department of Public Health(2020).
- [Background] Sorveglianza Integrata COVID-19 in Italia. Instituto Superiore di Sanitahttps://portale.fnomceo.it/wp-content/uploads/2020/04/Infografica_9aprile-ITA.pdf (2020).
- [Background] O'Donnell VB, Thomas D, Stanton R, Maillard JY, Murphy RC, Jones SA, Humphreys I, Wakelam MJO, Fegan C, Wise MP, Bosch A, Sattar SA. Potential Role of Oral Rinses Targeting the Viral Lipid Envelope in SARS-CoV-2 Infection. Function (Oxf). 2020;1(1):zqaa002. doi: 10.1093/function/zqaa002. Epub 2020 Jun 5. PMID 33215159
- [Background] Harrel SK, Molinari J. Aerosols and splatter in dentistry: a brief review of the literature and infection control implications. J Am Dent Assoc. 2004 Apr;135(4):429-37. doi: 10.14219/jada.archive.2004.0207. PMID 15127864
- [Background] Izzetti R, Nisi M, Gabriele M, Graziani F. COVID-19 Transmission in Dental Practice: Brief Review of Preventive Measures in Italy. J Dent Res. 2020 Aug;99(9):1030-1038. doi: 10.1177/0022034520920580. Epub 2020 Apr 17. PMID 32302257
- [Background] Ather A, Patel B, Ruparel NB, Diogenes A, Hargreaves KM. Reply to "Coronavirus Disease 19 (COVID-19): Implications for Clinical Dental Care". J Endod. 2020 Sep;46(9):1342. doi: 10.1016/j.joen.2020.08.005. Epub 2020 Aug 15. No abstract available. PMID 32810475
- [Background] Baghizadeh Fini M. What dentists need to know about COVID-19. Oral Oncol. 2020 Jun;105:104741. doi: 10.1016/j.oraloncology.2020.104741. Epub 2020 Apr 28. PMID 32380453
- [Background] Cleveland JL, Gray SK, Harte JA, Robison VA, Moorman AC, Gooch BF. Transmission of blood-borne pathogens in US dental health care settings: 2016 update. J Am Dent Assoc. 2016 Sep;147(9):729-38. doi: 10.1016/j.adaj.2016.03.020. Epub 2016 May 24. PMID 27233680
- [Background] Pfefferle, S. et al.Low and high infection dose transmission of SARS-CoV-2 in the first COVID-19 clusters in Northern Germany. medRxiv (2020) doi:10.1101/2020.06.11.20127332
- [Background] Ge ZY, Yang LM, Xia JJ, Fu XH, Zhang YZ. Possible aerosol transmission of COVID-19 and special precautions in dentistry. J Zhejiang Univ Sci B. 2020 May;21(5):361-368. doi: 10.1631/jzus.B2010010. Epub 2020 Mar 16. PMID 32425001
- [Background] Carrouel F, Conte MP, Fisher J, Goncalves LS, Dussart C, Llodra JC, Bourgeois D. COVID-19: A Recommendation to Examine the Effect of Mouthrinses with beta-Cyclodextrin Combined with Citrox in Preventing Infection and Progression. J Clin Med. 2020 Apr 15;9(4):1126. doi: 10.3390/jcm9041126. PMID 32326426
- [Background] Dennison DK, Meredith GM, Shillitoe EJ, Caffesse RG. The antiviral spectrum of Listerine antiseptic. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1995 Apr;79(4):442-8. doi: 10.1016/s1079-2104(05)80124-6. PMID 7614202
- [Background] Hasheminia D, Moaddabi A, Moradi S, Soltani P, Moannaei M, Issazadeh M. The efficacy of 1% Betadine mouthwash on the incidence of dry socket after mandibular third molar surgery. J Clin Exp Dent. 2018 May 1;10(5):e445-e449. doi: 10.4317/jced.54444. eCollection 2018 May. PMID 29849968
- [Background] Challacombe SJ, Kirk-Bayley J, Sunkaraneni VS, Combes J. Povidone iodine. Br Dent J. 2020 May;228(9):656-657. doi: 10.1038/s41415-020-1589-4. No abstract available. PMID 32385428
- [Background] Kirk-Bayley, J., Challacombe, S., Sunkaraneni, V. & Combes, J. The Use of Povidone Iodine Nasal Spray and Mouthwash During the Current COVID-19 Pandemic May Protect Healthcare Workers and Reduce Cross Infection. SSRN Electron. J.(2020) doi:10.2139/ssrn.3563092
- [Background] Statkute, E., Rubina, A., O'Donnell, V., Thomas, D., & Stanton, R. The Virucidal Efficacy of Oral Rinse Components Against SARS-CoV-2 In Vitro. BiorXiv. doi.org/10.1101/2020.11.13.381079
- [Background] COVID-19 Frequently Asked Questions. American Dental Association: Center for Professional Success (2020).
- [Background] Meiller TF, Silva A, Ferreira SM, Jabra-Rizk MA, Kelley JI, DePaola LG. Efficacy of Listerine Antiseptic in reducing viral contamination of saliva. J Clin Periodontol. 2005 Apr;32(4):341-6. doi: 10.1111/j.1600-051X.2005.00673.x. PMID 15811049
- [Background] Chapple ILC, Mealey BL, Van Dyke TE, Bartold PM, Dommisch H, Eickholz P, Geisinger ML, Genco RJ, Glogauer M, Goldstein M, Griffin TJ, Holmstrup P, Johnson GK, Kapila Y, Lang NP, Meyle J, Murakami S, Plemons J, Romito GA, Shapira L, Tatakis DN, Teughels W, Trombelli L, Walter C, Wimmer G, Xenoudi P, Yoshie H. Periodontal health and gingival diseases and conditions on an intact and a reduced periodontium: Consensus report of workgroup 1 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S74-S84. doi: 10.1002/JPER.17-0719. PMID 29926944
- [Background] Eke PI, Page RC, Wei L, Thornton-Evans G, Genco RJ. Update of the case definitions for population-based surveillance of periodontitis. J Periodontol. 2012 Dec;83(12):1449-54. doi: 10.1902/jop.2012.110664. Epub 2012 Mar 16. PMID 22420873

RESULTS

PARTICIPANT FLOW:
Groups:
- Peroxyl & Periogard: Subject participants will complete an on-label sequential rinse starting with Peroxyl (1.5% w/v hydrogen peroxide) 10 mL for 60 seconds and then Periogard (0.12% Chlorhexidine Gluconate) 15 mL for 30 seconds
- Colgate Total Zero: Subject participants will rinse mouth one time with Colgate Total Zero Fresh Breath (0.075% Cetylpyridinium Chloride) 20 mL for 30 seconds
Period: Overall Study
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
Started | 0 | 1 | 0 | 0 | 1
Completed | 0 | 1 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated after enrollment of only 2 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero | Total
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 0 | 0 | 1 | 2
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 1 | 2
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 1 | 0 | 0 | 1 | 2
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Reverse Transcription Polymerase Chain Reaction (RT-PCR) Baseline to 15 Min
Description: Determination of (RT-PCR) of inactivity of SARS-CoV-2 cellular infectivity in COVID+ patient saliva
Time Frame: Baseline, 15 minutes
Population: Due to early termination of the study, the biospecimen samples were destroyed and never analyzed.
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Change in Reverse Transcription Polymerase Chain Reaction (RT-PCR) From Baseline to 30 Minutes
Description: Determination of (RT-PCR) of inactivity of SARS-CoV-2 cellular infectivity in COVID+ patient saliva
Time Frame: Baseline, 30 Minutes
Population: Due to early termination of the study, the biospecimen samples were destroyed and never analyzed.
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Change in Reverse Transcription Polymerase Chain Reaction (RT-PCR) From Baseline to 45 Minutes
Description: Determination of (RT-PCR) of inactivity of SARS-CoV-2 cellular infectivity in COVID+ patient
Time Frame: Baseline, 45 Minutes
Population: Due to early termination of the study, the biospecimen samples were destroyed and never analyzed.
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Change in Reverse Transcription Polymerase Chain Reaction (RT-PCR) From Baseline to 60 Minutes
Description: Determination of (RT-PCR) of inactivity of SARS-CoV-2 cellular infectivity in COVID+ patient
Time Frame: Baseline, 60 minutes
Population: Due to early termination of the study, the biospecimen samples were destroyed and never analyzed.
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Change in Reverse Transcription Polymerase Chain Reaction (RT-PCR) From Baseline to 1-week.
Description: Determination of (RT-PCR) of inactivity of SARS-CoV-2 cellular infectivity in COVID+ patient
Time Frame: Baseline, 1 week
Population: Due to early termination of the study, the biospecimen samples were destroyed and never analyzed.
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change in Saliva Cytokine Concentration
Description: Change in inflammation-associated cytokine concentration (pg/mL) in saliva
Time Frame: Baseline, 1 week
Population: Due to early termination of the study, the biospecimen samples were destroyed and never analyzed.
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Change in Blood Cytokine Concentration
Description: Change in inflammation-associated cytokine concentration (pg/mL) in Blood
Time Frame: Baseline, 1 week
Population: Due to early termination of the study, the biospecimen samples were destroyed and never analyzed.
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Change in Saliva Chemokine Concentration
Description: Change in inflammation-associated chemokine concentration (pg/mL) in saliva
Time Frame: Baseline, 1 week
Population: Due to early termination of the study, the biospecimen samples were destroyed and never analyzed.
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Change in Blood Chemokine Concentration
Description: Change in inflammation-associated chemokine concentration (pg/mL) in Blood
Time Frame: Baseline, 1 week
Population: Due to early termination of the study, the biospecimen samples were destroyed and never analyzed.
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the signing of informed consent through the last visit, a total of approximately 1 week.
Description: Study terminated after enrollment of only 2 participants.
Arm/Group | Sterile Water | Peroxyl | Periogard | Peroxyl & Periogard | Colgate Total Zero
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT04748783/Prot_SAP_000.pdf